CLINICAL TRIAL: NCT06312397
Title: The Effect on Back Pain and Fatigue Level of Acupressure After Coronary Angiography: A Randomized, Single-Blind Sham-Controlled Study
Brief Title: The Effect on Back Pain and Fatigue Level of Acupressure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Birgul Vural Dogru, Associate Professor, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MU-HF-BVD-01
Record Dates: First submitted 2024-03-06; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Coronary Angiography
Keywords: Coronary angiography; Acupressure; Low back pain; Fatigue, Muscle
MeSH Terms: conditions — Low Back Pain; Fatigue | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: Three groups ( acupressure group, sham acupressure group and control group)
Who Masked: Participant
Masking Description: Patients in the acupressure and sham acupressure groups were blinded as to which groups they were in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupressure group (Active Comparator): After coronary angiography, acupressure will be applied for a total of 15 minutes. For the acupressure group, a total of three points will be applied: the heart meridian 7th point (HT7), the large intestine meridian 4th point (LI4), and the stomach meridian 36th point (ST36), which is deemed appropriate in the lower extremity.
  The symmetry of the three selected different points will also be applied to the other extremity.
  Interventions: Other: Acupressure
- Sham acupressure (Placebo Comparator): In the acupressure application applied to the sham group, parallel pressure will be applied to the bone area and points where the HT7, LI4, ST36 meridians do not pass.
  Interventions: Other: Sham acupressure
- Control group (No Intervention): With the control group, no intervention was conducted, and only standard care was given.

INTERVENTIONS:
Other: Acupressure — For the acupressure group, a total of three points will be applied: the heart meridian 7th point (HT7), the large intestine meridian 4th point (LI4), and the stomach meridian 36th point (ST36), which is deemed appropriate in the lower extremity The symmetry of the three selected different points will also be applied to the other extremity.
  After coronary angiography, acupressure will be applied for a total of 15 minutes.
  Arms: Acupressure group
Other: Sham acupressure — In the acupressure application applied to the sham group, parallel pressure will be applied to the bone area and points where the HT7, LI4, ST36 meridians do not pass.
  Arms: Sham acupressure

SUMMARY:
This research was conducted with the aim of determining the effect of acupressure on the level of back pain and fatigue after coronary angiography.

DETAILED DESCRIPTION:
To prevent bleeding, hematoma, and embolism after coronary angiography, patients are asked to stay in bed for 6 to 24 hours. During complete bed rest for at least 6 hours, the patient should keep his/her feet flat. The patient should lie in the supine position and avoid rapid movements. Long-term bed rest (at least 6 hours) in post-angiographic patients causes weakening of the lower back muscles and fatigue due to the pressure constantly applied to the same muscles, while muscle fatigue causes muscle spasms and lower back pain. Today, acupressure is also used along with various pharmacological treatments to relieve pain and fatigue.

Acupressure is a massage technique that ensures the proper functioning of energy channels by applying some pressure to certain parts of the body with the thumbs or index fingers, hands, palms, wrists and knees for therapeutic purposes. Acupressure points are the same as acupuncture points. Although there is no needle inserted into the body as in acupuncture.

According to G-power analysis, the total number of samples was calculated as 120.

A total of 120 participants will be randomly assigned to the acupuncture group (n=40), sham acupuncture group (n=40) and control group (n=40).

A Personal Information Form and Visual Analog Scales for Pain and Fatigue will be used to collect data.

ELIGIBILITY:
Inclusion Criteria:

* Planned coronary angiography from the femoral region
* Not diagnosed with low back pain
* No stent or other interventional procedure was performed during the coronary angiography procedure.

Exclusion Criteria:

* Those who have had acupressure before for any purpose
* Problems such as bleeding and dysrhythmia occur after coronary angiography,
* Those with burns, scars, scratches and deformities at the acupressure point
* Having any psychological disorder,

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale for Pain | 1 year
  It is used to measure subjectively perceived pain. On the scale, which includes the numbers between 0 and 10 cm, which are the most commonly used to determine the intensity of pain quantitatively, with painlessness at one end and the most severe pain possible at the other end, "0" defines painlessness and "10" defines the most severe pain.
Visual Analog Scale for Fatigue | 1 year
  The fatigue scale is a 10 cm scale that evaluates the severity of fatigue ranked from 0 to 10.
  On the left side of the scale, there is a rating of "I do not feel tired", and on the right side, there is a rating of "I feel extreme fatigue and exhaustion".

CONTACTS AND LOCATIONS:
Locations (1):
- Birgül VURAL DOĞRU, Mersin, Turkey (Türkiye)